CLINICAL TRIAL: NCT06035315
Title: The 1000 First Day of Life : Effect of Multi Micronutrients Supplementation on Pregnancy Outcomes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dr Cipto Mangunkusumo General Hospital (Other)
Responsible Party: Principal Investigator, Rima Irwinda, MD, OBGYN, PhD, Dr Cipto Mangunkusumo General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 23-02-0259
Record Dates: First submitted 2023-09-06; First posted 2023-09-13 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Maternal Care Patterns; Nutrition, Healthy; Nutritional Deficiency; Maternal-Fetal Relations; Perinatal Outcome; Maternal Outcome
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Intervention Model Description: Randomized control trial : comparison of two clusters
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (No Intervention): Pregnant women examine since 8 weeks gestation are being followed until delivery; are given government micronutrients; and perform ultrasound examinations each trimester and regular laboratory examination.
- Interventions (Active Comparator): Pregnant women examine since 8 weeks gestation are being followed until delivery; are given additional micronutrients (Complete multi micronutrients-Calcium-Vitamin D-DHA); and perform ultrasound examinations each trimester and additional laboratory examination (Vitamin D level-Lipid profile-Zinc)
  Interventions: Dietary Supplement: Multiple Micronutrients during pregnancy

INTERVENTIONS:
Dietary Supplement: Multiple Micronutrients during pregnancy — Pregnant women examine since 8 weeks gestation are being followed until delivery; are given additional micronutrients (Complete multi micronutrients-Calcium-Vitamin D-DHA); and perform ultrasound examinations each trimester and additional laboratory examination (Vitamin D level-Lipid profile-Zinc)
  Arms: Interventions

SUMMARY:
To monitor the effects of multi micronutrients supplementations during pregnancy towards pregnancy outcomes

DETAILED DESCRIPTION:
A randomized control trial of two clusters :

1st cluster without giving multi micronutrients; 2nd cluster giving multi micronutrients.

Differences between cluster : Additional multi micronutrients by giving : Complete multi micronutrients, calcium, vitamin D and DHA. The additional multi micronutrients were given since 1st until 3rd trimester for interventions group. There are also additional laboratory examinations for intervention group : Vitamin D, Lipid Profile and Zinc level.

In control group : we use standard public health care micronutrients (Iron supplementation and calcium); and standard blood examinations.

Ultrasound examination was performed for both cluster since 1st until 3rd trimester.

ELIGIBILITY:
Inclusion Criteria:

* First trimester pregnancy
* Gestational age < 10 weeks gestation
* Agree as research participant
* Living in DKI Jakarta

Exclusion Criteria:

* Assisted Reproductive
* History of PCOS
* History of Chronic Hypertension
* History of Diabetes Mellitus
* History of Preeclampsia
* Maternal chronic disease : Cardiovascular disease; Autoimmune condition; Malignancy)
* Plan to move from Jakarta prior or during pregnancy
* History of Recurrent pregnancy loss

Ages: 15 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 240 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Maternal Outcome | 1 year
  Maternal Death; Preterm Delivery; Preeclampsia; Intrauterine Infections; Post partum hemorrhage
Perinatal Outcome | 1 year
  Neonatal death; Low birth weight; Intra uterine growth restriction; Asphyxia

CONTACTS AND LOCATIONS:
Locations (2):
- Indonesia (2):
  - Cipto Mangunkusumo General Hospital, Jakarta Pusat, DKI Jakarta
  - Cipto Mangunkusumo General Hospital, Jakarta

IPD SHARING:
Plan to Share IPD: No